CLINICAL TRIAL: NCT05499507
Title: The Path to Optimal Black Maternal Heart Health: Comparing Two CVD Risk Reduction Interventions (Change of HEART)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27919
Record Dates: First submitted 2022-07-06; First posted 2022-08-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Hypertension; Obesity; Racism
MeSH Terms: conditions — Hypertension; Obesity; Racism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Change of Heart (COH) (Active Comparator): Incorporates two, evidence-based individual-level interventions (home blood pressure telemonitoring coupled with the interactive obesity treatment approach, that includes nutrition and physical activity text messages with tailored feedback) and an institutional-level intervention (anti-racism training of providers and staff along with patient feedback to inform respectful care).
  Interventions: Behavioral: COH
- Change of Heart Plus (COH+) (Experimental): Includes all components of COH plus the addition of interpersonal support for Black women by Black women (community doula care, mental health services, and lactation support).
  Interventions: Behavioral: COH+

INTERVENTIONS:
Behavioral: COH — Incorporates two, evidence-based individual-level interventions (home blood pressure telemonitoring coupled with the interactive obesity treatment approach, that includes nutrition and physical activity text messages with tailored feedback) and an institutional-level intervention (anti-racism training of providers and staff along with patient feedback to inform respectful care).
  Arms: Change of Heart (COH)
Behavioral: COH+ — Includes all components of COH plus interpersonal support for Black women by Black women (community doula care, mental health services, and lactation support).
  Arms: Change of Heart Plus (COH+)

SUMMARY:
The overarching goal of our proposal is to reduce disparities in perinatal cardiovascular disease risk factors among Black women utilizing a community-driven, social ecological framework.

DETAILED DESCRIPTION:
What is this research about? Heart disease (e.g., heart attack, stroke) is a major threat to safe motherhood and is the leading cause of maternal death in the United States, responsible for nearly 50 percent of pregnancy-related deaths among Black women, three times the rate of white women, and is largely preventable. It is well established that eating healthy foods and monitoring blood pressure can help prevent heart disease. While prior studies addressing these individual behaviors have led to some success, a single individual-level approach has not been enough to stop the rising rate of Black maternal mortality. Researchers have also established that depression, social isolation, and stress from racism lead to poor heart outcomes. But few studies have treated these psychosocial and structural factors in addition to individual behaviors to ensure optimal Black maternal heart health, particularly for mothers at higher risk (e.g., those with high blood pressure and/or obesity). To meet this need, the research team plans to compare two approaches that treat multiple factors leading to heart disease among 432 patients age 18 and older who self-identify as Black or African American, have either obesity and/or high blood pressure, are less than 24 weeks pregnant, and have a smart phone. Both approaches address individual behaviors through nutrition and physical activity text messages and home blood pressure self-monitoring as well as provide training to medical care providers in order to reduce patients' experiences of racism or mistreatment. But only one of the approaches being studied also adds supports for Black women by Black women (community doula care, mental health services, and lactation consultation) during their pregnancy, birth, and postpartum in order to learn if these supports lead to lower blood pressure and also treat social isolation, depression, and increase experiences of respectful maternity care.

Who can this research help? This study will increase Black mothers' understanding of the many influences on their heart health. Findings from this study will help Black women with obesity and/or high blood pressure make informed decisions about the use of community doulas, lactation professionals, and psychotherapists as part of their care to reduce risks for heart disease during pregnancy or in the first year after their baby is born. Results may also strengthen health systems' commitment to anti-racism training as part of their efforts to provide quality health care for Black pregnant and postpartum people. And further, this research may provide evidence to insurance companies that coverage of this study's package of supports is needed.

What outcomes are being studied? The primary outcomes are changes in maternal blood pressure and body weight at six weeks and one year after giving birth. The team will also evaluate how well the treatments are implemented and able to reach patients, be adopted into practice consistently, and lead to healthcare provider and patient satisfaction. The team will analyze outcomes that patient partners have identified as important. These include perinatal mood and anxiety disorders (e.g., postpartum depression), emotional and informational support, stress, and experiences of respectful maternity care. In addition, the study team will look at clinical outcomes including if and for how long patients breastfeed, blood pressure disorders of pregnancy, how the patient gave birth (e.g., vaginal or cesarean), baby's birth weight, and how many weeks pregnant mothers were at the time of birth.

How long does this study last? Final follow-up of primary outcomes is at one year postpartum (i.e., approximately 18 months from enrollment).

How are stakeholders involved? The research team believes that efforts to improve Black maternal heart health will be most effective when partnered with patients and community leaders that have shared lived experience. Study leadership is an equitable partnership by an academic physician-researcher and community-based Black provider who herself experienced heart health complications in her pregnancy. There are three other patient investigators who will also be involved in all aspects of the planning, delivery, and evaluation of the treatments, including serving as lead doulas, therapists, and lactation professionals. Patient representatives will make up the majority of the study's advisory board to give feedback and further guide the team's efforts throughout the five years of the project. Finally, patient, health system, and community provider stakeholders will provide feedback and guidance through focus groups over the entire study duration to ensure adoption of treatments.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* baseline BMI ≥30 kg/m2 and/or diagnosis of HTN (≥130/80 x 2)
* gestational age <24 weeks by last menstrual period
* smartphone ownership
* self-identification as Black or African American

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure at 6-weeks postpartum. | At baseline and 6-weeks postpartum
  Blood pressure will be measured at each time point on the upper arm three times at one-minute intervals after five minutes of quiet sitting. The investigators will use the validated Omron HEM-907XL and the appropriate size cuff. The investigators will average the three measures for analysis.
Change in blood pressure at 12-months postpartum. | At baseline and 12-months postpartum
  Blood pressure will be measured at each time point on the upper arm three times at one-minute intervals after five minutes of quiet sitting. The investigators will use the validated Omron HEM-907XL and the appropriate size cuff. The investigators will average the three measures for analysis.
Change in body weight at 6-weeks postpartum. | At baseline and 6-weeks postpartum
  Body weight will be measured in duplicate and recorded to the nearest 0.1kg using calibrated SECA scales at each time point.
Change in body weight at 12-months postpartum. | At baseline and 12-months postpartum
  Body weight will be measured in duplicate and recorded to the nearest 0.1kg using calibrated SECA scales at each time point.

SECONDARY OUTCOMES:
Change in emotional support at 6-weeks postpartum. | At baseline and 6-weeks postpartum
  The investigators will use the 8-item emotional support PROMIS instrument to measure perceived feelings of being cared for at each time point. The lowest possible raw score is 8; the highest possible raw score is 40. Higher scores indicate greater emotional support.
Change in emotional support at 12-months postpartum. | At baseline and 12-months postpartum
  The investigators will use the 8-item emotional support PROMIS instrument to measure perceived feelings of being cared for at each time point. The lowest possible raw score is 8; the highest possible raw score is 40. Higher scores indicate greater emotional support.
Change in informational support at 6-weeks postpartum. | At baseline and 6-weeks postpartum
  The investigators will use the 8-item informational support PROMIS instruments to measure perceived availability of helpful information or advice at each time point. The lowest possible raw score is 8; the highest possible raw score is 40. Higher scores indicate greater informational support.
Change in informational support at 12-months postpartum. | At baseline and 12-months postpartum
  The investigators will use the 8-item informational support PROMIS instruments to measure perceived availability of helpful information or advice at each time point. The lowest possible raw score is 8; the highest possible raw score is 40. Higher scores indicate greater informational support.
Change in Perinatal Mood and Anxiety Disorders (PMADs) at 6-weeks postpartum. | At baseline and 6-weeks postpartum
  PMADs will be assessed using the Beck Depression Inventory II (BDI-II), a 21-item screening tool. The BDI-II has demonstrated concurrent validity with other postpartum depression scales and validated cut points for mild/moderate depressive symptoms in Black women of low-socioeconomic position. The lowest possible raw score is 1; the highest possible raw score is 40. Higher scores indicate greater depressive symptoms.
Change in PMADs at 12-months postpartum. | At baseline and 12-months postpartum
  PMADs will be assessed using the Beck Depression Inventory II (BDI-II), a 21-item screening tool. The BDI-II has demonstrated concurrent validity with other postpartum depression scales and validated cut points for mild/moderate depressive symptoms in Black women of low-socioeconomic position. The lowest possible raw score is 1; the highest possible raw score is 40. Higher scores indicate greater depressive symptoms.
Mothers autonomy in decision making at baseline. | Baseline
  The 7-item Mothers Autonomy in Decision Making scale rates patients' level of agency and autonomy experienced during conversations with a maternity provider. The range of scores is 7-42, with higher scores indicating more opportunities to take an active role and lead decisions.
Mothers autonomy in decision making at 6-weeks postpartum. | 6-weeks postpartum
  The 7-item Mothers Autonomy in Decision Making scale rates patients' level of agency and autonomy experienced during conversations with a maternity provider. The range of scores is 7-42, with higher scores indicating more opportunities to take an active role and lead decisions.
Respectful maternity care at baseline. | Baseline
  Respectful maternity care will be assessed by the 14-item Mothers on Respect Index, which examines the nature of provider-patient relationships and access to person-centered care. The range of scores is 14-84, with higher scores indicating more respectful care.
  lead decisions.
Respectful maternity care at 6-weeks postpartum. | 6-weeks postpartum
  Respectful maternity care will be assessed by the 14-item Mothers on Respect Index, which examines the nature of provider-patient relationships and access to person-centered care. The range of scores is 14-84, with higher scores indicating more respectful care.
Obstetric mistreatment at baseline. | Baseline
  The 8-item Mistreatment Index queries patients' experience of dimensions of mistreatment (e.g., physical abuse, discrimination). To describe the overall prevalence of mistreatment, the investigators will calculate the proportion of women who experienced each of the seven types of mistreatment and what proportion experience any mistreatment (i.e. any of the seven indicators).
Obstetric mistreatment at 6-weeks postpartum | 6-weeks postpartum
  The 8-item Mistreatment Index queries patients' experience of dimensions of mistreatment (e.g., physical abuse, discrimination). To describe the overall prevalence of mistreatment, the investigators will calculate the proportion of women who experienced each of the seven types of mistreatment and what proportion experience any mistreatment (i.e. any of the seven indicators).
Blood pressure control at 6-weeks postpartum for patients with hypertension (HTN) at baseline. | 6-weeks postpartum
  Blood pressure control will be assessed at each time point for patients with HTN at enrollment (proportion with mean systolic BP ≥ 130mm/Hg or mean diastolic BP ≥ 80mm/Hg).
Blood pressure control at 12-months postpartum for patients with hypertension at baseline. | 12-months postpartum
  Blood pressure control will be assessed at each time point for patients with HTN at enrollment (proportion with mean systolic BP ≥ 130mm/Hg or mean diastolic BP ≥ 80mm/Hg).
Incident hypertension at 6-weeks postpartum for patients who were normotensive at baseline. | 6-weeks postpartum
  Data will be collected about incident HTN at 6-weeks and 1-year postpartum for normotensive patients at enrollment (proportion with mean systolic BP ≥130 mm/Hg or mean diastolic BP ≥ 80mm/Hg).
Incident hypertension at 12-months postpartum for patients who were normotensive at baseline. | 12-months postpartum
  Data will be collected about incident HTN at 6-weeks and 1-year postpartum for normotensive patients at enrollment (proportion with mean systolic BP ≥130 mm/Hg or mean diastolic BP ≥ 80mm/Hg).
Breast/Chestfeeding initiation. | 6-weeks postpartum
  Breast/chestfeeding initiation will be assessed via questions adapted from the Infant Feeding Practices Study II.
Breast/Chestfeeding duration. | 12-months postpartum
  Breast/chestfeeding duration will be assessed via questions adapted from the Infant Feeding Practices Study II.
Breastfeeding support/self-efficacy at 6-weeks postpartum. | 6-weeks postpartum
  Breast/chestfeeding self-efficacy will be assessed via questions adapted from the Breastfeeding Self-Efficacy Scale. The range of scores is 14-70, with higher scores indicating greater self-efficacy.
Breastfeeding support/self-efficacy at 12-months postpartum. | 12-months postpartum
  Breast/chestfeeding self-efficacy will be assessed via questions adapted from the Breastfeeding Self-Efficacy Scale. he range of scores is 14-70, with higher scores indicating greater self-efficacy.
Mode of delivery. | 6-weeks postpartum
  Mode of delivery will be abstracted from the electronic health record and categorized as either operative delivery (cesarean section) or non-operative (vaginal delivery), stratified by birth history.
Infant birth weight. | 6-weeks postpartum
  Infant birth weight will be abstracted from electronic health record. The investigators will calculate sex-specific birth weight for gestational age percentile based on national data.
Preterm birth. | 6-weeks postpartum
  To determine rates of preterm birth, gestational length will be calculated from last menstrual period (LMP) unless ultrasound dating differs ≥10 days from LMP dating. Pregnancy loss will be assessed by self-report, verified by electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon J Herring, MD, MPH, Principal Investigator — Temple University, Philadelphia, Pennsylvania, United States, 19140
Locations (1):
- Temple University/Temple Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Descriptions of the study dataset, including codebooks and documentation of the programming code used for creating the final study population, variable definitions, and descriptive and outcome analyses will be provided at the end of the final funding year. The investigators will make these materials, as well as the final dataset, available via the Inter-university Consortium for Political and Social Research (ICPSR, https://www.icpsr.umich.edu/web/pages/) of which Temple University is a member.
Time Frame: 8/10/2027

REFERENCES:
- [Derived] Wycoff KL, Coleman JG, Santoro CM, Zullig LL, Darden N, Holland PM, Cruice JF, Mitchell S, Smith M, McNeil SJ, Herring SJ. Multilevel Community Engagement to Inform a Randomized Clinical Trial. Obstet Gynecol. 2023 Oct 1;142(4):929-939. doi: 10.1097/AOG.0000000000005344. Epub 2023 Sep 7. PMID 37734093